CLINICAL TRIAL: NCT07368348
Title: Evaluation of Internal Nasal Splint-Supported Free Graft Versus Nasoseptal Flap for Endoscopic Skull Base Repair in Cerebrospinal Fluid Leaks
Acronym: CSF
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Kafrelsheikh University (Other)
Collaborators: Faculty of medicine kafr elshiekh university (Unknown)
Responsible Party: Principal Investigator, Amr Mahr Shady, resident, Kafrelsheikh University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: KFSIRB200-695
Record Dates: First submitted 2025-12-25; First posted 2026-01-26 (Actual); Last update posted 2026-01-26 (Actual); Status verified 2025-09

CONDITIONS: CSF Leak
Keywords: CSF, Stent
MeSH Terms: conditions — Cerebrospinal Fluid Otorrhea

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Nasoseptal Flap for Endoscopic Skull (Experimental): • Group A: Free graft + Internal nasal splint
  * Free graft material (e.g., fascia lata, fat, synthetic dural substitute) placed over the defect.
  * Internal nasal splint applied to support the graft and maintain its position
  Interventions: Device: Nasoseptal Flap for Endoscopic Skull Base Repair in Cerebrospinal Fluid Leaks
- Evaluation of Internal Nasal Splint-Supported Free Graft in Endoscopic Skul (Experimental): • Group B: Nasoseptal flap alone.
  - Standard nasoseptal flap technique used for skull base repair.
  Interventions: Device: Internal Nasal Splint-Supported Free Graft

INTERVENTIONS:
Device: Internal Nasal Splint-Supported Free Graft — Evaluation of Internal Nasal Splint-Supported Free Graft versus Nasoseptal Flap for Endoscopic Skull Base Repair in Cerebrospinal Fluid Leaks
  Arms: Evaluation of Internal Nasal Splint-Supported Free Graft in Endoscopic Skul
Device: Nasoseptal Flap for Endoscopic Skull Base Repair in Cerebrospinal Fluid Leaks — Nasoseptal Flap for Endoscopic Skull Base Repair in Cerebrospinal Fluid Leaks
  Arms: Nasoseptal Flap for Endoscopic Skull

SUMMARY:
The study aims to compare the feasibility and effectiveness of using an internal nasal splint- supported free graft versus a nasoseptal flap alone for endoscopic repair of bilateral CSF leaks.

Research question:

Does the use of an internal nasal splint to support a free graft during endoscopic repair of bilateral CSF leaks improve outcomes compared to the use of a nasoseptal flap alone?

DETAILED DESCRIPTION:
Cerebrospinal fluid (CSF) leaks are classified as traumatic, iatrogenic, or spontaneous/idiopathic. Traumatic causes include blunt or penetrating facial injuries, while iatrogenic causes stem from neurosurgical or otolaryngologic procedures, such as Functional Endoscopic Sinus Surgery (FESS).

Spontaneous CSF leaks, often linked to elevated intracranial pressure (ICP), may occur in conditions like Idiopathic Intracranial Hypertension (IIH) or due to congenital skull base defects and tumors [2]. Risk factors for spontaneous leaks include obesity, female gender, and obstructive sleep apnea, with studies showing 72% of affected patients are female and 45% have sleep apnea.

Benign Intracranial Hypertension (BIH), also known as IIH or Pseudotumor Cerebri (PTC), involves increased brain pressure without structural abnormalities and normal CSF content. Spontaneous CSF rhinorrhea, increasingly prevalent (14-55%), often requires thorough investigations (e.g., fundus examination, CT/MRI, neurological consultation) to exclude intracranial hypertension before endoscopic repair.

Lumbar drain with CSF manometry is reserved for recurrent cases, often due to benign CSF tension increases despite normal preoperative findings. Successful repair requires competent flaps/grafts to withstand CSF pressure during healing. Recurrence necessitates further investigations and may require additional CSF diversion or shunting.

Key steps for successful repair include:

1. Identifying the defect(s).
2. Creating a raw area around the defect by removing mucosa.
3. Precisely placing a graft or flap, optionally sealing dural tears with fat or fascia.
4. Applying adequate pressure to counteract CSF pressure.

Sealing mechanisms involve:

1. Tucking a graft or fat under bony edges or into dural tears, though this may risk dural trauma.
2. Applying a free graft or vascularized flap over the defect and surrounding bone, requiring pressure equal to or greater than CSF pressure. Combining both mechanisms with adequate pressure optimizes sealing and compensates for potential weaknesses.

From a physical perspective, grafts or flaps must exert force equal to or greater than CSF pressure to prevent leaks. On-lay grafts require sufficient force, while under-lay grafts, though challenging, benefit from additional on-lay grafts or flaps to address unnoticed defects.

Nasoseptal flaps (NSFs) have become a widely used technique for endoscopic skull base repair, particularly for cerebrospinal fluid (CSF) leaks. They are vascularized pedicled flaps that provide a robust and reliable option for sealing skull base defects. Studies have shown that NSFs have high success rates, ranging from 90% to 95%, in preventing CSF leaks postoperatively. The vascularity of the flap promotes healing and reduces the risk of graft failure, making it a preferred choice for large or complex defect.

However, NSFs are not without limitations. The technique requires a relatively intact nasal septum, which may not be feasible in patients with prior septal surgery, large septal perforations, or severe septal deformities. Additionally, harvesting the flap can lead to complications such as nasal crusting, septal perforation, and nasal obstruction, which can affect patient quality of life.

Free grafts, such as fascia lata, fat, or synthetic dural substitutes, are another option for skull base repair. These grafts are non-vascularized and rely on the surrounding tissue for nourishment. Free grafts are simpler to harvest and place, making them a viable option in cases where NSFs are not feasible. However, their success rates are generally lower than those of NSFs, with reported success rates ranging from 70% to 85%.

The main challenge with free grafts is their susceptibility to displacement and failure due to the pressure exerted by CSF. Without adequate support, free grafts may not adhere properly to the defect, leading to recurrent leaks. Techniques to improve the stability of free grafts, such as the use of fibrin glue or additional support materials, have been explored, but these methods have not consistently improved outcomes.

The study aims to evaluate the effectiveness of internal nasal splints in improving the feasibility and success rate of free grafts during endoscopic CSF leak repair.

ELIGIBILITY:
Inclusion Criteria: 1- Adults (≥18 years). 2- Patients with bilateral CSF leaks confirmed by imaging and biochemical testing (e.g., beta-2 transferrin).

3- Patients with bilateral CSF leak and sever septal spur. 4- Patients with bilateral CSF leak and history of submucosal resection of nasal septum.

5- Patients with bilateral CSF leak and large septal perforation. 6- Patients with bilateral CSF Leak and septal granuloma.

Exclusion Criteria: 1- Patients with contraindications to endoscopic surgery. 2- Active sinus or nasal infections. 3- Previous nasal or skull base surgery affecting the repair site.

-

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2026-02-01 (Estimated); Primary Completion 2026-06-01 (Estimated); Study Completion 2026-11-01 (Estimated)

PRIMARY OUTCOMES:
Evaluation of Internal Nasal Splint-Supported Free Graft versus Nasoseptal Flap for Endoscopic Skull Base Repair in Cerebrospinal Fluid Leaks | baseline
  • Primary Objective:
  - To evaluate the effectiveness of internal nasal splints in improving the feasibility and success rate of free grafts during endoscopic repair of bilateral CSF leaks.

CONTACTS AND LOCATIONS:
Locations (1):
- Kafrelsheikh Faculty of Medicine, Kafr Elsheikh, Kafrelsheikh, Egypt

IPD SHARING:
Plan to Share IPD: Undecided
anyone who is interestd in this study.

REFERENCES:
- [Result] Kim-Orden N, Shen J, Or M, Hur K, Zada G, Wrobel B. Endoscopic Endonasal Repair of Spontaneous Cerebrospinal Fluid Leaks Using Multilayer Composite Graft and Vascularized Pedicled Nasoseptal Flap Technique. Allergy Rhinol (Providence). 2019 Nov 13;10:2152656719888622. doi: 10.1177/2152656719888622. eCollection 2019 Jan-Dec. PMID 31763054